CLINICAL TRIAL: NCT05519644
Title: Strategies to Augment Ketosis: Ketone Conferred Resiliency Against Sleep Restriction
Acronym: STAK-Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jeff Volek, Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022H0169; CDMRP-PR212399-C (Other Grant/Funding Number: Departent of Defense)
Record Dates: First submitted 2022-08-18; First posted 2022-08-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation | interventions — Heart Rate; Diet; Surveys and Questionnaires; Reaction Time; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: A double-blind, placebo-controlled, two-period cross-over study
Who Masked: Participant, Investigator
Masking Description: Study product will be distributed in a blinded manner by people not involved with testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo First (Active Comparator): Patients will be randomize to take the placebo for the first trial of the intervention, then after a 2 week washout, participants will perform the same intervention but with a ketone ester.
  Interventions: Other: Sleep Deprivation; Other: Heart Rate; Other: Sleep Monitoring; Other: Diet; Other: Exercise Performance; Behavioral: Surveys, McGill Pain Questionnaire, Shortened Profile of Mood States, Pittsburg Sleep Index; Other: Cognitive performance; Other: Marksmanship Performance; Other: Quick Board; Other: Advanced Medical Technologies Inc, Jump Test; Other: CGM/CKM; Biological: Blood Draw; Dietary Supplement: Ketone Supplement
- Ketone Ester First (Experimental): Patients will be randomize to take the ketone ester for the first trial of the intervention, then after a 2 week washout, participants will perform the same intervention but with a placebo
  Interventions: Other: Sleep Deprivation; Other: Heart Rate; Other: Sleep Monitoring; Other: Diet; Other: Exercise Performance; Behavioral: Surveys, McGill Pain Questionnaire, Shortened Profile of Mood States, Pittsburg Sleep Index; Other: Cognitive performance; Other: Marksmanship Performance; Other: Quick Board; Other: Advanced Medical Technologies Inc, Jump Test; Other: CGM/CKM; Biological: Blood Draw; Dietary Supplement: Ketone Supplement

INTERVENTIONS:
Other: Sleep Deprivation — The sleeping protocol will be monitored by investigators and personnel with experience in sleep medicine. Participants will be required to reduce sleep by 50% of normal, for 4 consecutive nights, to observe potential deficits in physical and cognitive performance
Other: Heart Rate — HR will be assessed by wrist-based acceleration with cloud technology (Polar Unite™, Polar USA). This monitor is less burdensome than other sleep monitoring technologies and less likely to interfere with normal sleep and activity demands of the cadets. Each participant will be fitted with the watch for acclimatization and then establish 3-day baseline patterns for 3 nights before the sleep loss protocol.
Other: Sleep Monitoring — Sleep will be assessed by wrist-based acceleration with cloud technology (Polar Unite™, Polar USA). This monitor is less burdensome than other sleep monitoring technologies and less likely to interfere with normal sleep and activity demands of the cadets.Each participant will be fitted with the watch for acclimatization and then establish 3-day baseline patterns for 3 nights before the sleep loss protocol.
Other: Diet — Diet will be included and the same meals will be available for all subjects while controlling for caffeine. Participants will be given food during each intervention week.
Other: Exercise Performance — Since weight training is now a crucial part of any warfighter's physical preparation, we will have subjects perform weight training workouts emphasizing all major muscle groups on Days 2, 3 and 4
Behavioral: Surveys, McGill Pain Questionnaire, Shortened Profile of Mood States, Pittsburg Sleep Index — These will be administered on Days 1 and 5 of each intervention trial to assess different behavioral outcomes.
Other: Cognitive performance — Automated Neuropsychological Assessment Metrics (ANAM), Cambridge Neuropsychological Test Automated Battery. (CANTAB),Gradual-onset Continuous Performance Task (GRAD-CPT),Face-Name Task will be used to assess cognitive function and performance.
Other: Marksmanship Performance — The Virtual Training Simulator (VirTra V-100) system (VirTra Corporate HQ, Tempe, AZ) is used by both military and law enforcement agencies to provide training. The V-100 and associated compatible weapons are equipped with recoil kits for unsurpassed live-fire simulation, at distances up to 2,000-m, authoring capabilities for the creation of customized scenarios on 4 individual firing lanes. Multiple metrics of marksmanship (total number of shots fired/silhouette target presentation, percentage of targets successfully hit/min, the radial distance of a shot from the center on target, shot group tightness, and time from target presentation to trigger pull) will be collected during each visit.
  Other Names: VirTra
Other: Quick Board — Upper body and lower body reaction tests will be assess using Quick Board Analysis on days 1 and 5 of the sleep restriction intervention.
  Other Names: Response Time
Other: Advanced Medical Technologies Inc, Jump Test — Whole body power will be assessed with a repetitive jump test. Power (peak, average, curve functions) will be assessed using an AMTI force plate with Accupower 2.0 software (Advanced Mechanical Technology Inc, Watertown, MA).
  Other Names: Whole Body Power
Other: CGM/CKM — Continuous Ketone/Glucose Monitor will be applied at the start of Test Day 1. The sensor will be checked by the study team at each test day and will be removed and replaced by a fresh sensor at ~2- week intervals during the study. The sensor will be removed at the end of the final test day.
Biological: Blood Draw — Blood samples will be collected according to the schedule in Figure 1.
Dietary Supplement: Ketone Supplement — Participants will take a diester of hexanoic acid (a ketogenic medium chain fatty acid) and (R)-1,3 butanediol (C6 Di-ester) during one of the trial interventions

SUMMARY:
Sleep deprivation is a major problem in military populations. Some major consequences of sleep loss are inability to concentrate, poor work efficiency, and increase in errors during daily tasks. There is some evidence that ketone ester supplements may lessen the adverse effects of sleep restriction. The main purpose of these supplements is to raise your blood concentration of ketones, which are safe, small molecules that appear in the blood during fasting, when following a ketogenic diet, or consuming ketone supplements.

The main purpose of this study is to examine if ingesting a ketone ester supplement, twice daily, can improve cognitive and physical performance during short-term sleep restriction.

DETAILED DESCRIPTION:
Only 1 in 3 U.S. Army Active Component Soldiers are estimated to get the target =7-hr of sleep on duty days, and ~14% have a sleep disorder. Insufficient sleep has profound effects on human performance that include deficits in working memory, creativity, innovative thinking, strategic planning, mood disturbances, lapses in attention and vigilance, and impaired physical performance. In a classic dose-response sleep study performed at Walter Reed Army Institute of Research, it was demonstrated that limiting sleep to 3-hr per night for 7-days resulted in a steady deterioration on a psychomotor vigilance task across the week of sleep restriction. Sleep restriction over 3-days has been shown to adversely affect marksmanship performance, including significantly longer time to make decisions, misidentifying friends versus foes, and believing performance did not change over time. Short-term sleep restriction is linked with impaired glucose metabolism and decreased whole body insulin sensitivity, and increases the risk of developing T2D. Military personnel have few good options to counteract physical and cognitive detriments attributed to insufficient sleep. Warfighters increasingly turn to caffeine and sugar-containing energy drinks to combat sleep loss and fatigue, especially during deployment. At best, these nutritional countermeasures provide a transient performance gain, and may trigger a 'rebound' hypoglycemia that exacerbates performance detriments that can increase the risk of obesity and related problems. Ketosis could improve tolerance to sleep restriction and sleep abnormalities through multiple mechanisms. We have reported that a 1-yr KD improved sleep quality and the proportion of people categorized as poor sleepers. Ketones are a preferred brain fuel that may enhance neurocognitive function. The ability to metabolize a lipid-derived substrate (ketones) capable of sustaining the brain's high energy demands during periods with limited access to carbohydrate was a central adaptation in human evolution, that is also associated with a remarkable protection from the adverse signs of hypoglycemia. At the low end of nutritional ketosis (0.5 mM), ~5% of whole brain energy metabolism is provided by ketones. At ketone concentrations of 1.5 mM (typical of KDs), ketones supply nearly 20%; at the higher end of nutritional ketosis 4-5 mM [achievable with ketone esters (KE)], half of the brain energy demands are met by ketones. Importantly in situations where brain glucose metabolism is impaired, uptake and utilization of ketones remain fully intact, suggesting a hierarchy of importance placed on ketones as the preferred fuel for human brains.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to comply with all study procedures including the following prior to Test Days: fasting (>10 h; water only), no alcohol (>24 h), no exercise (>24 h), no acute illness and controlled feeding before each Test Day, maintain diet, exercise, medication, and supplement habits throughout the study.
* Participant has no health conditions that would prevent completion of the study requirements as judged by the Investigator based on health history.
* Participant understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Investigator.

Exclusion Criteria:

* <18 or >40 years of age
* >35 body mass index (BMI).
* Diagnosed sleeping disorders (i.e., sleep apnea, insomnia).
* Gastrointestinal disorders or food allergies that would interfere with consuming the study supplements.
* Drink alcohol in excess of 3 drinks/day or 14 drinks/week
* Have any conditions or contraindications to blood draws.
* Have been diagnosed with diabetes, liver, kidney, or other metabolic or endocrine dysfunction, or use diabetic medications other than metformin
* Currently consume a low carbohydrate or ketogenic diet or have done so in the last 3 months
* Have experienced weight loss of >10% of your body weight within the last 6 months
* Are pregnant, lactating, or planning on becoming pregnant during the study
* Have any major psychiatric disorders (e.g., schizophrenia, bipolar disorder)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Automated Neuropsychological Assessment Metrics (ANAM) | Up to ~ 4 weeks
  This cognitive battery is a library of computer-based tests of domains including attention, concentration, reaction time, memory, processing speed, decision-making, and executive function.
Cambridge Neuropsychological Test Automated Battery. (CANTAB) | Up to ~ 4 Weeks
  This iPad delivery assessment will include an Information Sampling Task to test impulsivity and decision making, response time (in msec), which provides a level of sensitivity not available with traditional paper and pencil tasks, processing speed, executive functioning, and spatial memory. We have also incorporated tasks which assess the ability to rapidly identify expressed facial emotions, which may index one's ability to accurately respond to overtly threatening or non-threatening stimuli
Gradual-onset Continuous Performance Task (GRAD-CPT | Up to ~4 weeks
  This test measures endogenous attentional control by using smooth (rather than abrupt) transitions between visual images. Scene stimuli are visually presented and smoothly transition from one scene to another. Subjects press a button when one type of scene is presented (e.g., city scene) and withhold the button press when another type of scene (e.g., mountain scene) is presented. It is a Go/No-Go test and assesses multiple metrics of executive function, including sustained attention, mind wandering, and response inhibition.
Face-Name Task | Up to ~4 weeks
  We will implement a face-name relational memory task, known to activate the hippocampus (along with prefrontal and parietal cortices) in humans using face-name pairs presented for 3-sec with an interval of 750-msec. Participants will judge which name was previously presented with the face. After a 15-min delay, participants will complete an associative face-name recognition task to assess episodic memory performance.
Total number of shots fired | Up to ~4 weeks
  The Virtual Training Simulator (VirTra V-100) system (VirTra Corporate HQ, Tempe, AZ) is used by both military and law enforcement agencies to provide training. The V-100 and associated compatible weapons are equipped with recoil kits for unsurpassed live-fire simulation, at distances up to 2,000-m, authoring capabilities for the creation of customized scenarios on 4 individual firing lanes. Total number of shots fired, a metric of marksmanship, will be collected during each visit, to assess reaction time and accuracy.
Percentage of targets successfully hit per minute | Up to ~4 weeks
  The Virtual Training Simulator (VirTra V-100) system (VirTra Corporate HQ, Tempe, AZ) is used by both military and law enforcement agencies to provide training. The V-100 and associated compatible weapons are equipped with recoil kits for unsurpassed live-fire simulation, at distances up to 2,000-m, authoring capabilities for the creation of customized scenarios on 4 individual firing lanes. Percentage of targets successfully hit/min, a metric of marksmanship, will be collected during each visit to assess accuracy.
Radial distance of a shot from the center on target | Up to ~4 weeks
  The Virtual Training Simulator (VirTra V-100) system (VirTra Corporate HQ, Tempe, AZ) is used by both military and law enforcement agencies to provide training. The V-100 and associated compatible weapons are equipped with recoil kits for unsurpassed live-fire simulation, at distances up to 2,000-m, authoring capabilities for the creation of customized scenarios on 4 individual firing lanes. The radial distance of a shot from the center on target, a metric of marksmanship, will be collected during each visit to assess shot accuracy.
Shot Group Tightness | Up to ~4 weeks
  The Virtual Training Simulator (VirTra V-100) system (VirTra Corporate HQ, Tempe, AZ) is used by both military and law enforcement agencies to provide training. The V-100 and associated compatible weapons are equipped with recoil kits for unsurpassed live-fire simulation, at distances up to 2,000-m, authoring capabilities for the creation of customized scenarios on 4 individual firing lanes. Shot group tightness, a metric of marksmanship, will be collected during each visit to assess multi-shot accuracy.
Time from target presentation to trigger pull | Up to ~4 weeks
  The Virtual Training Simulator (VirTra V-100) system (VirTra Corporate HQ, Tempe, AZ) is used by both military and law enforcement agencies to provide training. The V-100 and associated compatible weapons are equipped with recoil kits for unsurpassed live-fire simulation, at distances up to 2,000-m, authoring capabilities for the creation of customized scenarios on 4 individual firing lanes. Time from target presentation to trigger pull, a metric of marksmanship , will be collected during each visit to assess reaction time.
Power Outcome (QuickBoard) | Up to ~4 weeks
  Upper body and lower body reaction tests will be assess using Quick Board Analysis on days 1 and 5 of the sleep restriction intervention.

SECONDARY OUTCOMES:
CGM/CKM | Up to ~ 4 weeks
  Diurnal concentrations of ketones and glucose via a continuous monitor. The ketone sensor in this CKM device is similar to the FreeStyle Libre continuous glucose monitoring (CGM). The sensor adheres to the back of the arm where it continuously samples interstitial fluid for quantification of BHB concentration. The sensor is worn for a period of 2-wk, two sensors will be used to cover all test days in this study (4 weeks including 2 week washout)
Heart Rate | Up to ~ 4 weeks
  HR will be assessed by wrist-based acceleration with cloud technology (Polar Unite™, Polar USA). This will allow for assessment of changes in HR.
Short Form- McGill Pain Questionnaire | Up to ~ 4 weeks
  The Short Form McGill pain questionnaire (SF-MPQ) will be used to assess pain in individuals. Clinically important change (CIC): mean improvement in total scores >5 on the 0-45 SF-MPQ scale. Minimum detectable change (MDC) for total, sensory, affective, average, and current pain: 5.2cm, 4.5cm, 2.8cm, 1.4cm, and 1.4cm, respectively. The SF-MPQ will be examined around the sleep restriction/exercise intervention on Days 1 and 5 to assess pain change.
Profile of Mood States- Short Form | Up to ~ 4 weeks
  Shortened Profile of Mood States- Short Form (POMS-SF) measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment. For each word and statement, they must circle the number on a Likert scale from 0= Not at all to 4=Extremely for how often they have felt those feelings today and over the past week. The POMS-SF will be examined around the sleep restriction/exercise intervention on Days 1 and 5 to assess mood.
Pittsburgh Sleep Quality Index | Up to ~ 4 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. PSQI will be examined around the sleep restriction/exercise intervention on Days 1 and 5 to assess sleep quality.
Insulin | Up to ~ 4 weeks
  Differences in blood hormones insulin after supplementation will be analyzed using commercially available ELISA assay kits (Cayman Chemical, USA).
Ghrelin | Up to ~ 4 weeks
  Differences in blood hormones insulin after supplementation will be analyzed using commercially available ELISA assay kits (Cayman Chemical, USA).
CRP | Up to ~ 4 weeks
  Differences in blood proteins after supplementation will be analyzed using commercially available ELISA assay kits (Cayman Chemical, USA).
Brain Derived Neurotropic Factor | Up to ~4 weeks
  Differences in neurotrophins after supplementation will be analyzed using commercially available ELISA assay kits (Cayman Chemical, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S Volek, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: OSU Office of Responsible Research Practices — http://orrp.osu.edu

DOCUMENTS (2):
  • Study Protocol (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT05519644/Prot_000.pdf
  • Informed Consent Form (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT05519644/ICF_001.pdf